CLINICAL TRIAL: NCT07010302
Title: A Comparative Clinical Effectiveness Trial of Rituximab Versus Ravulizumab, Inebilizumab, Satralizumab and Eculizumab To Prevent Relapses in Neuromyelitis Optica Spectrum Disorder
Brief Title: Rituximab Versus Ravulizumab, Inebilizumab, Satralizumab, and Eculizumab in NMOSD
Acronym: BEST-NMOSD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Charite University, Berlin, Germany (Other); The Sumaira Foundation (Unknown)
Responsible Party: Principal Investigator, Philippe A. Bilodeau, MD, Principal investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 40200
Record Dates: First submitted 2025-05-21; First posted 2025-06-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: NMOSD
MeSH Terms: interventions — Rituximab; eculizumab; ravulizumab; satralizumab; inebilizumab

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Rituximab (Active Comparator)
  Interventions: Drug: Rituximab (R)
- Complement inhibitors (Experimental): Ravulizumab or eculizumab
  Interventions: Drug: Eculizumab (Soliris®); Drug: Ravulizumab
- Inebilizumab (Experimental)
  Interventions: Drug: Inebilizumab
- Satralizumab (Experimental)
  Interventions: Drug: Satralizumab
- Open-label, non-randomized (Other): Open-label, non-randomized
  Interventions: Drug: Rituximab (R); Drug: Eculizumab (Soliris®); Drug: Ravulizumab; Drug: Satralizumab; Drug: Inebilizumab

INTERVENTIONS:
Drug: Rituximab (R) — 1000 mg at weeks 0 and 2 followed by 1000 mg every 6 months
  Other Names: Rituxan; Truxima
  Arms: Open-label, non-randomized; Rituximab
Drug: Eculizumab (Soliris®) — 900 mg weekly for 4 weeks, followed by 1200 mg every 2 weeks
  Arms: Complement inhibitors; Open-label, non-randomized
Drug: Ravulizumab — * 40 to < 60 kg: 2400 mg
  * 60 to < 100 kg: 2700 mg
  * 100 kg: 3000 mg as an induction dose, followed by
  * 40 to < 60 kg: 3000 mg
  * 60 to < 100 kg: 3300 mg
  * 100 kg: 3600 mg Every 8 weeks starting 15 days after loading dose
  Arms: Complement inhibitors; Open-label, non-randomized
Drug: Satralizumab — 120 mg at Weeks 0, 2, 4, followed by 120 mg every 4 weeks
  Arms: Open-label, non-randomized; Satralizumab
Drug: Inebilizumab — 300 mg on Day 1 and Day 15, followed by 300 mg every 6 months
  Arms: Inebilizumab; Open-label, non-randomized

SUMMARY:
Neuromyelitis Optica Spectrum Disorder (NMOSD) is a rare autoimmune condition that mainly affects the eyes and spinal cord, causing serious symptoms such as vision loss, paralysis, and severe pain. This trial compares the effectiveness and safety of five medications commonly used to prevent NMOSD relapses: rituximab, ravulizumab, inebilizumab, satralizumab, and eculizumab.

In this study, 160 adults with NMOSD who test positive for a specific antibody (AQP4-IgG) will participate. They will be randomly assigned to receive either rituximab or one of the four other FDA-approved medications. The main goal is to find out which treatment best prevents relapses and has fewer serious side effects. The trial will also measure disability, patient satisfaction, quality of life, and biomarkers that help track disease activity.

Participants will have regular assessments, including medical exams, surveys, and tests for vision, walking ability, and brain function. They will report any side effects or health issues experienced during the study. The trial will last from one to four years for each participant.

This research aims to help patients and doctors make better-informed treatment decisions by providing clear evidence about the best available therapies for NMOSD.

DETAILED DESCRIPTION:
Neuromyelitis Optica Spectrum Disorder (NMOSD) is an autoimmune inflammatory disorder primarily affecting the optic nerves and spinal cord, leading to symptoms such as blindness, severe muscle weakness, paralysis, and significant pain. This study aims to directly compare the clinical effectiveness and safety profiles of five distinct therapies widely utilized to prevent disease relapses in patients with NMOSD who test positive for aquaporin-4 antibodies (AQP4-IgG): rituximab, ravulizumab, inebilizumab, satralizumab, and eculizumab.

The study is designed as an international, multicenter, randomized, adaptive clinical trial. It involves enrolling 160 adult participants diagnosed with AQP4-IgG positive NMOSD, who will be randomized in equal numbers to receive either rituximab or one of the four other FDA-approved therapies-ravulizumab, inebilizumab, satralizumab, or eculizumab. Patients randomized to the non-rituximab group will undergo further randomization into one of these four comparator medications. Additionally, the study incorporates an observational cohort for patients who decline randomization but agree to be followed according to the same protocol.

The primary objective is to evaluate the comparative effectiveness of rituximab versus the other treatments in preventing NMOSD relapses and treatment failure due to adverse events. Secondary objectives include comparing disability outcomes, evaluating treatment-related adverse events, and assessing impacts on patient-reported quality of life, as well as examining changes in biomarkers relevant to NMOSD disease activity.

Participants will undergo comprehensive evaluations at regular intervals, including detailed neurological examinations, standardized functional assessments (Expanded Disability Status Scale [EDSS], Multiple Sclerosis Functional Composite [MSFC]), visual acuity and contrast sensitivity testing, and cognitive assessments. Additionally, patient-reported outcomes such as fatigue, pain, mental health status, and overall quality of life will be collected systematically through validated surveys. Safety assessments will include regular monitoring of blood work, clinical evaluations for infections and other complications, and documentation of all adverse events.

Advanced exploratory analyses will also include biomarker studies involving optical coherence tomography (OCT) to assess retinal nerve fiber layer loss, and assays for serum neurofilament light chain (NfL) and glial fibrillary acidic protein (GFAP) levels. The study will track direct and indirect healthcare costs, as well as impacts on employment and caregiver burden.

The duration of participation will range from one to four years, depending on when participants enroll and their clinical outcomes. All data will be rigorously analyzed using advanced statistical methods, including time-to-event analyses, mixed-effects models, and Bayesian hierarchical approaches to allow robust comparative effectiveness evaluations.

Ultimately, this research aims to provide high-quality, head-to-head data to inform clinical decision-making, optimize treatment strategies, and improve patient outcomes for those living with NMOSD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NMOSD according to the 2015 International Panel for NMO Diagnosis (IPND) consensus criteria.
* Seropositivity for AQP4 immunoglobulin G (AQP4-IgG) confirmed by a cell-based assay (either live or fixed) that meets the threshold for positivity set by the local testing laboratory.
* Age ≥18 years at the time of consent.
* Ability and willingness to provide informed consent and comply with all study procedures, including scheduled visits, laboratory tests, and assessments.
* Eligible to receive any of the study drugs based on clinical judgment

Exclusion Criteria:

* Known active hepatitis B virus (HBV) infection, defined as a positive hepatitis B surface antigen or detectable HBV DNA by PCR.
* Known active hepatitis C virus (HCV) infection, defined as detectable HCV RNA by PCR.
* Known active or latent tuberculosis, evidenced by a positive interferon-gamma release assay (IGRA) unless fully treated per local guidelines before enrollment.
* Known or suspected immunodeficiency disorders, including but not limited to HIV infection with CD4 count <200 cells/mm³ or any condition requiring chronic immunosuppressive therapy outside the scope of the study drugs.
* Pregnancy or breastfeeding, or intention to conceive during the study period. Pregnancy is excluded due to insufficient safety data for the investigational treatments in this population. Women of childbearing potential must agree to use effective contraception throughout the study and for a defined period following the last dose of study drug, per product labeling or institutional guidance.
* Any medical, psychiatric, or neurological condition that, in the investigator's opinion, may interfere with study participation, pose additional risk to the participant, or confound interpretation of study results.
* Inability or unwillingness to comply with the requirements of the protocol, including scheduled visits, evaluations, or procedures, based on investigator assessment.
* Known hypersensitivity or severe allergic reaction to any component of the study drugs or pre-medications required for infusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Time to adjudicated safety or tolerability failure | From date of randomization until the date of first adjudicated safety or tolerability failure or adjudicated relapse, whichever comes first, assessed up to 48 months
  Includes adverse events, tolerability, patient preference, or logistical barriers.
Time to adjudicated relapse | From date of randomization until the date of adjudicated relapse or first treatment discontinuation, whichever comes first, assessed up to 48 months
  As determined by the blinded Relapse Adjudication Committee using pre-specified clinical and imaging criteria

SECONDARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | Baseline and every 12 months through study completion, an average of 30 months and a maximum of 48 months
  Quantifies the severity of disability in patients with neuroinflammatory disorders such as NMOSD. The scale ranges from 0 to 10 in half-point increments, where 0 indicates normal neurological function and 10 represents death due to neurological causes. Higher scores reflect greater disability.
Timed 25-Foot Walk | Baseline and every 12 months through study completion, an average of 30 months and a maximum of 48 months
  Measures ambulatory function. Participants are instructed to walk 25 feet as quickly and safely as possible. The time to complete the walk is recorded; lower times indicate better function.
9-Hole Peg Test | Baseline and every 12 months through study completion, an average of 30 months and a maximum of 48 months
  Assesses upper extremity function and fine motor coordination. Participants place and remove nine pegs into a pegboard as quickly as possible using one hand. The test is performed separately for each hand. The time to complete the task is recorded; shorter times reflect better performance.
Symbol Digit Modalities Test (SDMT) | Baseline and every 12 months through study completion, an average of 30 months and a maximum of 48 months
  Evaluates cognitive processing speed. Participants are presented with a series of symbols matched with numbers and asked to substitute the corresponding number for each symbol within 90 seconds. The total number of correct responses is recorded; higher scores indicate better cognitive performance.
Landolt High Contrast Visual Acuity | Baseline and every 12 months through study completion, an average of 30 months and a maximum of 48 months
  Assessed using Landolt ring optotypes under standard lighting conditions. Participants identify the orientation of the ring (gap in one of four cardinal directions). The number of correct responses is converted to a visual
Landolt Low Contrast Visual Acuity | Baseline and every 12 months through study completion, an average of 30 months and a maximum of 48 months
  Assessed using Landolt ring optotypes at 2.5% contrast. Participants identify the orientation of the ring (gap in one of four cardinal directions). The number of correct responses is converted to a visual acuity ratio (Snellen equivalent). Higher ratios indicate better low contrast vision.
Treatment Satisfaction Questionnaire for Medication II (TSQM-II) | Baseline and every 6 months through study completion, an average of 30 months and a maximum of 48 months
  Assesses patient satisfaction with medication across multiple domains, including effectiveness, side effects, convenience, and global satisfaction. Higher scores indicate greater satisfaction with treatment.
EuroQol 5-Dimension 5-Level (EQ-5D-5L) | Baseline and every 6 months through study completion, an average of 30 months and a maximum of 48 months
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression . Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. Index values, calculated using country-specific value sets, range from less than 0 (health states considered worse than death) to 1 (full health). An associated visual analog scale (VAS) records the respondent's self-rated health on a scale from 0 (worst imaginable health) to 100 (best imaginable health).
PROMIS Depression Short form | Baseline and every 6 months through study completion, an average of 30 months and a maximum of 48 months
  8-item self-report questionnaire used to assess depression
Fatigue Scale for Motor and Cognitive Function | Baseline and every 6 months through study completion, an average of 30 months and a maximum of 48 months
  20-item patient-reported measure assessing both motor and cognitive fatigue in individuals with neuroinflammatory diseases. It yields separate subscale scores and a total fatigue score; higher scores indicate greater fatigue.
Visual Function Questionnaire 25 | Baseline and every 6 months through study completion, an average of 30 months and a maximum of 48 months
  Neasures vision-related quality of life across 12 subscales, including general vision, ocular pain, and social functioning. It is designed for individuals with chronic eye diseases. Higher scores indicate better self-reported visual function.
Brief Pain Inventory | Baseline and every 6 months through study completion, an average of 30 months and a maximum of 48 months
  Evaluates pain severity and the impact of pain on daily functions. It includes both numeric rating scales and interference items related to activity, mood, walking, and sleep. Higher scores on severity and interference scales indicate more severe and impactful pain.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe-Antoine Bilodeau, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barreras P, Vasileiou ES, Filippatou AG, Fitzgerald KC, Levy M, Pardo CA, Newsome SD, Mowry EM, Calabresi PA, Sotirchos ES. Long-term Effectiveness and Safety of Rituximab in Neuromyelitis Optica Spectrum Disorder and MOG Antibody Disease. Neurology. 2022 Nov 29;99(22):e2504-e2516. doi: 10.1212/WNL.0000000000201260. Epub 2022 Aug 31. PMID 36240094
- [Background] Yamamura T, Weinshenker B, Yeaman MR, De Seze J, Patti F, Lobo P, von Budingen HC, Kou X, Weber K, Greenberg B. Long-term safety of satralizumab in neuromyelitis optica spectrum disorder (NMOSD) from SAkuraSky and SAkuraStar. Mult Scler Relat Disord. 2022 Oct;66:104025. doi: 10.1016/j.msard.2022.104025. Epub 2022 Jul 5. PMID 36007339
- [Background] Rensel M, Zabeti A, Mealy MA, Cimbora D, She D, Drappa J, Katz E. Long-term efficacy and safety of inebilizumab in neuromyelitis optica spectrum disorder: Analysis of aquaporin-4-immunoglobulin G-seropositive participants taking inebilizumab for ⩾4 years in the N-MOmentum trial. Mult Scler. 2022 May;28(6):925-932. doi: 10.1177/13524585211047223. Epub 2021 Oct 1. PMID 34595983
- [Background] Kumpfel T, Giglhuber K, Aktas O, Ayzenberg I, Bellmann-Strobl J, Haussler V, Havla J, Hellwig K, Hummert MW, Jarius S, Kleiter I, Klotz L, Krumbholz M, Paul F, Ringelstein M, Ruprecht K, Senel M, Stellmann JP, Bergh FT, Trebst C, Tumani H, Warnke C, Wildemann B, Berthele A; Neuromyelitis Optica Study Group (NEMOS). Update on the diagnosis and treatment of neuromyelitis optica spectrum disorders (NMOSD) - revised recommendations of the Neuromyelitis Optica Study Group (NEMOS). Part II: Attack therapy and long-term management. J Neurol. 2024 Jan;271(1):141-176. doi: 10.1007/s00415-023-11910-z. Epub 2023 Sep 7. PMID 37676297
- [Background] Nosadini M, Alper G, Riney CJ, Benson LA, Mohammad SS, Ramanathan S, Nolan M, Appleton R, Leventer RJ, Deiva K, Brilot F, Gorman MP, Waldman AT, Banwell B, Dale RC. Rituximab monitoring and redosing in pediatric neuromyelitis optica spectrum disorder. Neurol Neuroimmunol Neuroinflamm. 2016 Jan 21;3(1):e188. doi: 10.1212/NXI.0000000000000188. eCollection 2016 Feb. PMID 26819962
- [Background] Rover C, Friede T. Dynamically borrowing strength from another study through shrinkage estimation. Stat Methods Med Res. 2020 Jan;29(1):293-308. doi: 10.1177/0962280219833079. Epub 2019 Mar 1. PMID 30821201
- [Background] Wingerchuk DM, Banwell B, Bennett JL, Cabre P, Carroll W, Chitnis T, de Seze J, Fujihara K, Greenberg B, Jacob A, Jarius S, Lana-Peixoto M, Levy M, Simon JH, Tenembaum S, Traboulsee AL, Waters P, Wellik KE, Weinshenker BG; International Panel for NMO Diagnosis. International consensus diagnostic criteria for neuromyelitis optica spectrum disorders. Neurology. 2015 Jul 14;85(2):177-89. doi: 10.1212/WNL.0000000000001729. Epub 2015 Jun 19. PMID 26092914
- [Background] Marcinno A, Marnetto F, Valentino P, Martire S, Balbo A, Drago A, Leto M, Capobianco M, Panzica G, Bertolotto A. Rituximab-induced hypogammaglobulinemia in patients with neuromyelitis optica spectrum disorders. Neurol Neuroimmunol Neuroinflamm. 2018 Sep 13;5(6):e498. doi: 10.1212/NXI.0000000000000498. eCollection 2018 Nov. PMID 30258855
- [Background] Clardy SL, Pittock SJ, Aktas O, Nakahara J, Isobe N, Centonze D, Fam S, Kielhorn A, Yu JC, Jansen J, Zhang I. Network Meta-analysis of Ravulizumab and Alternative Interventions for the Treatment of Neuromyelitis Optica Spectrum Disorder. Neurol Ther. 2024 Jun;13(3):535-549. doi: 10.1007/s40120-024-00597-7. Epub 2024 May 9. PMID 38722571
- [Background] Yamamura T, Kleiter I, Fujihara K, Palace J, Greenberg B, Zakrzewska-Pniewska B, Patti F, Tsai CP, Saiz A, Yamazaki H, Kawata Y, Wright P, De Seze J. Trial of Satralizumab in Neuromyelitis Optica Spectrum Disorder. N Engl J Med. 2019 Nov 28;381(22):2114-2124. doi: 10.1056/NEJMoa1901747. PMID 31774956
- [Background] Pittock SJ, Barnett M, Bennett JL, Berthele A, de Seze J, Levy M, Nakashima I, Oreja-Guevara C, Palace J, Paul F, Pozzilli C, Yountz M, Allen K, Mashhoon Y, Kim HJ. Ravulizumab in Aquaporin-4-Positive Neuromyelitis Optica Spectrum Disorder. Ann Neurol. 2023 Jun;93(6):1053-1068. doi: 10.1002/ana.26626. Epub 2023 Apr 5. PMID 36866852
- [Background] Pittock SJ, Berthele A, Fujihara K, Kim HJ, Levy M, Palace J, Nakashima I, Terzi M, Totolyan N, Viswanathan S, Wang KC, Pace A, Fujita KP, Armstrong R, Wingerchuk DM. Eculizumab in Aquaporin-4-Positive Neuromyelitis Optica Spectrum Disorder. N Engl J Med. 2019 Aug 15;381(7):614-625. doi: 10.1056/NEJMoa1900866. Epub 2019 May 3. PMID 31050279
- [Background] Tahara M, Oeda T, Okada K, Kiriyama T, Ochi K, Maruyama H, Fukaura H, Nomura K, Shimizu Y, Mori M, Nakashima I, Misu T, Umemura A, Yamamoto K, Sawada H. Safety and efficacy of rituximab in neuromyelitis optica spectrum disorders (RIN-1 study): a multicentre, randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2020 Apr;19(4):298-306. doi: 10.1016/S1474-4422(20)30066-1. Epub 2020 Mar 18. PMID 32199095
- [Background] Kim SH, Huh SY, Lee SJ, Joung A, Kim HJ. A 5-year follow-up of rituximab treatment in patients with neuromyelitis optica spectrum disorder. JAMA Neurol. 2013 Sep 1;70(9):1110-7. doi: 10.1001/jamaneurol.2013.3071. PMID 23897062
- [Background] Kleiter I, Gold R. Present and Future Therapies in Neuromyelitis Optica Spectrum Disorders. Neurotherapeutics. 2016 Jan;13(1):70-83. doi: 10.1007/s13311-015-0400-8. PMID 26597098
- [Background] Trebst C, Jarius S, Berthele A, Paul F, Schippling S, Wildemann B, Borisow N, Kleiter I, Aktas O, Kumpfel T; Neuromyelitis Optica Study Group (NEMOS). Update on the diagnosis and treatment of neuromyelitis optica: recommendations of the Neuromyelitis Optica Study Group (NEMOS). J Neurol. 2014 Jan;261(1):1-16. doi: 10.1007/s00415-013-7169-7. Epub 2013 Nov 23. PMID 24272588
- [Background] Sellner J, Boggild M, Clanet M, Hintzen RQ, Illes Z, Montalban X, Du Pasquier RA, Polman CH, Sorensen PS, Hemmer B. EFNS guidelines on diagnosis and management of neuromyelitis optica. Eur J Neurol. 2010 Aug;17(8):1019-32. doi: 10.1111/j.1468-1331.2010.03066.x. Epub 2010 Jun 7. PMID 20528913
- [Background] Mealy MA, Kessler RA, Rimler Z, Reid A, Totonis L, Cutter G, Kister I, Levy M. Mortality in neuromyelitis optica is strongly associated with African ancestry. Neurol Neuroimmunol Neuroinflamm. 2018 Jun 7;5(4):e468. doi: 10.1212/NXI.0000000000000468. eCollection 2018 Jul. No abstract available. PMID 29892608
- [Background] Kim SH, Mealy MA, Levy M, Schmidt F, Ruprecht K, Paul F, Ringelstein M, Aktas O, Hartung HP, Asgari N, Tsz-Ching JL, Siritho S, Prayoonwiwat N, Shin HJ, Hyun JW, Han M, Leite MI, Palace J, Kim HJ. Racial differences in neuromyelitis optica spectrum disorder. Neurology. 2018 Nov 27;91(22):e2089-e2099. doi: 10.1212/WNL.0000000000006574. Epub 2018 Oct 26. PMID 30366977
- [Background] Duchow A, Bellmann-Strobl J, Friede T, Aktas O, Angstwurm K, Ayzenberg I, Berthele A, Dawin E, Engels D, Fischer K, Flaskamp M, Giglhuber K, Grothe M, Havla J, Hummert MW, Jarius S, Kaste M, Kern P, Kleiter I, Klotz L, Korporal-Kuhnke M, Kraemer M, Krumbholz M, Kumpfel T, Lohmann L, Ringelstein M, Rommer P, Schindler P, Schubert C, Schwake C, Senel M, Then Bergh F, Tkachenko D, Tumani H, Trebst C, Vardakas I, Walter A, Warnke C, Weber MS, Wickel J, Wildemann B, Winkelmann A, Paul F, Stellmann JP, Haussler V; Neuromyelitis Optica Study Group (NEMOS). Time to Disability Milestones and Annualized Relapse Rates in NMOSD and MOGAD. Ann Neurol. 2024 Apr;95(4):720-732. doi: 10.1002/ana.26858. Epub 2024 Jan 13. PMID 38086777
- [Background] Kleiter I, Gahlen A, Borisow N, Fischer K, Wernecke KD, Wegner B, Hellwig K, Pache F, Ruprecht K, Havla J, Krumbholz M, Kumpfel T, Aktas O, Hartung HP, Ringelstein M, Geis C, Kleinschnitz C, Berthele A, Hemmer B, Angstwurm K, Stellmann JP, Schuster S, Stangel M, Lauda F, Tumani H, Mayer C, Zeltner L, Ziemann U, Linker R, Schwab M, Marziniak M, Then Bergh F, Hofstadt-van Oy U, Neuhaus O, Winkelmann A, Marouf W, Faiss J, Wildemann B, Paul F, Jarius S, Trebst C; Neuromyelitis Optica Study Group. Neuromyelitis optica: Evaluation of 871 attacks and 1,153 treatment courses. Ann Neurol. 2016 Feb;79(2):206-16. doi: 10.1002/ana.24554. Epub 2015 Nov 26. PMID 26537743
- [Background] O'Connell K, Hamilton-Shield A, Woodhall M, Messina S, Mariano R, Waters P, Ramdas S, Leite MI, Palace J. Prevalence and incidence of neuromyelitis optica spectrum disorder, aquaporin-4 antibody-positive NMOSD and MOG antibody-positive disease in Oxfordshire, UK. J Neurol Neurosurg Psychiatry. 2020 Oct;91(10):1126-1128. doi: 10.1136/jnnp-2020-323158. Epub 2020 Jun 23. No abstract available. PMID 32576617
- [Background] Briggs FB, Shaia J. Prevalence of neuromyelitis optica spectrum disorder in the United States. Mult Scler. 2024 Jan 27:13524585231224683. doi: 10.1177/13524585231224683. Online ahead of print. PMID 38279789
- [Background] Kitley J, Leite MI, Nakashima I, Waters P, McNeillis B, Brown R, Takai Y, Takahashi T, Misu T, Elsone L, Woodhall M, George J, Boggild M, Vincent A, Jacob A, Fujihara K, Palace J. Prognostic factors and disease course in aquaporin-4 antibody-positive patients with neuromyelitis optica spectrum disorder from the United Kingdom and Japan. Brain. 2012 Jun;135(Pt 6):1834-49. doi: 10.1093/brain/aws109. Epub 2012 May 9. PMID 22577216
- [Background] Haussler V, Trebst C, Engels D, Pellkofer H, Havla J, Duchow A, Schindler P, Schwake C, Pakeerathan T, Fischer K, Ringelstein M, Lindenblatt G, Hummert MW, Tkachenko D, Butow F, Giglhuber K, Flaskamp M, Schiffmann I, Korporal-Kuhnke M, Jarius S, Dawin E, Revie L, Senel M, Herfurth M, Walter A, Pompsch M, Kleiter I, Angstwurm K, Kaste M, Grothe M, Wickel J, Rommer PS, Sieb JP, Kramer M, Then Bergh F, Tumani H, Klotz L, Wildemann B, Aktas O, Ayzenberg I, Bellmann-Strobl J, Paul F, Kumpfel T, Friede T, Berthele A, Stellmann JP; Neuromyelitis optica study group (NEMOS). Real-world multicentre cohort study on choices and effectiveness of immunotherapies in NMOSD and MOGAD. J Neurol Neurosurg Psychiatry. 2025 May 14;96(6):582-592. doi: 10.1136/jnnp-2024-334764. PMID 39730197